CLINICAL TRIAL: NCT02976597
Title: Morphine as an Adjunct in Sonar Guided Transversus Abdominis Plane Block for Postoperative Analgesia in Patients Undergoing Abdominal Surgery.
Brief Title: Ultrasound Guided TAP Block for Postoperative Analgesia After Abdominal Surgery.
Acronym: TAB
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Assisstant professor in anesthesia and intensive care, Faculty of medicine, Assiut university, Egypt., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17100234
Record Dates: First submitted 2016-11-24; First posted 2016-11-29 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Postoperative Pain
Keywords: Abdominal surgery, pain, local, transversus abdominus block.
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Bupivacaine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bupivacaine 0.25% (Active Comparator): Bupivacaine 0.25% 20ml will be administered for ultrasound guided TAP block on each side on each side at end of the surgery.
  Interventions: Drug: Bupivacaine 0.25% 20ml on each side Sonar guided TAB
- Morphine 10mg (Active Comparator): Morphine 10mg and Bupivacaine 0.25% 20ml will be administered for ultrasound guided TAP block on each side at end of the surgery.Patients will recieve 5mg morphine on each side
  Interventions: Drug: Bupivacaine 0.25% 20ml on each side Sonar guided TAB; Drug: Morphine 10mg
- Morphine 15mg (Active Comparator): Morphine 15mg and Bupivacaine 0.25% 20ml will be administered for ultrasound guided TAP block on each side at end of the surgery. Patients will recieve 7.5mg morphine on each side
  Interventions: Drug: Bupivacaine 0.25% 20ml on each side Sonar guided TAB; Drug: Morphine 15mg

INTERVENTIONS:
Drug: Bupivacaine 0.25% 20ml on each side Sonar guided TAB — Bupivacaine 0.25% 20ml on each side Sonar guided TAP block. After careful aspiration injection of 20ml of 0.25% bupivacaine will be performed and hypoechoic layer will be detected on ultrasound then the maneuver will be repeated on the other side
  Other Names: BUCAIN Sonar guided
Drug: Morphine 10mg — Morphine 10mg will be added to bupivacaine in sonar guided- TAP block divided into 5mg on each side.
  Other Names: Morphine injection
  Arms: Morphine 10mg
Drug: Morphine 15mg — Morphine 15mg will be added to bupivacaine in sonar guided- TAP block divided into 7.5mg on each side.
  Other Names: Morphine injection
  Arms: Morphine 15mg

SUMMARY:
Transversus abdominis plane (TAP) block is a novel type of peripheral nerve block that involves innervations of the anterolateral abdominal wall derived from T6-L1.It provides adequate post-operative pain relieve following the various abdominal surgeries. Theoretically, TAP block may replace the need for epidural analgesia after abdominal operations. The oblique subcostal approach of the TAP (OSTAP) block, which was de¬scribed by (Hebbard et al, 2010) , has been reported to provide analgesia to the entire anterior abdomen.

DETAILED DESCRIPTION:
The transversus abdominis plane (TAP) technique, originally described by involves injection of local anaesthetic in the plane between the internal oblique and transversus abdominis muscle layers, with the aim of anaesthetising the intercostal nerves supplying the abdominal wall. Initially, the block used surface landmarks of the triangle of Petit (latissimus dorsi posteriorly, external oblique superiorly, iliac crest inferiorly) and a double fascial 'pop' (loss of resistance) to guide placement of the local anaesthetic. More recently, ultrasonography has been used to guide the delivery of the injectate into the appropriate plane, thereby increasing the accuracy of the Technique.

The duration of the TAB is limited to effect of administered local anesthetics. To prolong the block's duration, adjuvant medications were added to LA to magnify the effect of TAP block . Opiates such as morphine and tramadol have peripheral and central analgesic effects. Opiate receptors are present at the terminals of afferent peripheral nerves; therefore, administration of opiates peripherally might provide a significant analgesic effect.

ELIGIBILITY:
Inclusion Criteria:

BMI< 30kg/m2.

* Age: 18-60 years.
* Sex: both males and females.
* ASA physical status: 1-II.
* Operation: Abdominal laparotomy.

Exclusion Criteria:

* Patient refusal.
* History of cardiac disease, psychological disorders, respiratory diseases including asthma, renal or hepatic failure.
* Coagulation disorders.
* Allergy to study medications.
* Chronic use of pain medications.
* Pregnancy.
* Respiratory tract in-fection within the last 2 weeks.
* Heavy smoker.
* Histo-ry of abdominal surgery or trauma.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Verbal Rating Scale Score | 24 hours
  The 24 hours postoperative verbal rating scale score on cough

SECONDARY OUTCOMES:
Time to first request of rescue analgesia. | 24 hours
  The total 24 hours consumption of analgesic drugs taken.
Time to first request of rescue analgesics. | 24 hours
  The time from end of the operation, PACU admission and the request for analgesic drugs.
Spirometric assessment | 24 hours
  Measurment of lung function by spirometry.
Adverse effects | 24 hours
  Recording and treatment of adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Principal Investigator — Assisstant professor in anesthesia and intensive care, faculty of medicine, Assiut university, Egypt
Locations (1):
- Hala Saad Abdel-Ghaffar, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No